CLINICAL TRIAL: NCT06539013
Title: Efficacy of Remifentanil in Preventing Emergence Agitation in Patients Undergoing Nasal Surgery Under Desflurane Anesthesia: A Prospective Double-blind Randomized Controlled Trial.
Brief Title: Efficacy of Remifentanil in Preventing Emergence Agitation
Acronym: agitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTosunSONE
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Remifentanil; Analgesia; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 Remifentanily (Active Comparator): Patients in Group 1 received 0.05-0.2 μg/kg/min IV remifentanil infusion as analgesic.
  Interventions: Drug: Remifentanil
- group 2 N2O (Active Comparator): N2O instead of 50% air was applied to patients in Group 2 for intraoperative analgesia.
  Interventions: Drug: N2O
- group 3 Fentanly (Active Comparator): In addition to Desflurane, 50% oxygen and 50% air, 1 μg/kg IV fentanyl bolus was administered as analgesic when there was a 20% increase in heart rate and blood pressure values during the operation for patients in Group 3.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — remifentanil infusion
  Other Names: Use of remifentanil infusion for analgesia
  Arms: group 1 Remifentanily
Drug: N2O — Use of N2O for analgesia
  Other Names: Use of N2O for analgesia
  Arms: group 2 N2O
Drug: Fentanyl — Use of Fentanylfor analgesia
  Other Names: Use of Fentanyl for analgesia
  Arms: group 3 Fentanly

SUMMARY:
The primary aim of the study was to test the hypothesis that remifentanil administered for analgesia prevents emergence agitation more effectively than fentanyl and N2O in patients undergoing rhinoplasty who received desflurane as an inhaled anesthetic agent. The secondary aim of the study was to compare the demographic data, intraoperative and postoperative hemodynamic data, surgical time and modified Aldrete score of patients who received different intraoperative analgesia methods.

ELIGIBILITY:
Inclusion Criteria:

The study included patients over the age of 18, planned to undergo rhinoplasty by the plastic and reconstructive surgery department, and American Society of Anesthesiologist (ASA) I-II.

-

Exclusion Criteria:

* Patients with a known history of allergy to the drugs to be administered in the study, ASA III and above, body mass index (BMI) 35>kg/m2, younger than 18 years of age, any problems that would prevent general anesthesia in the preoperative evaluation (upper respiratory tract infection, etc.), and those who did not agree to participate in the study were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) | Postoperative care unit 1.second_5. second_15.second
  * 4 Combative, violent, danger to staff
  * 3 Pulls or removes tube(s) or catheters; aggressive
  * 2 Frequent non-purposeful movement, fights ventilator
  * 1 Anxious, apprehensive, but not aggressive 0 Alert and calm
    * 1 Awakens to voice (eye opening/contact) > 10 seconds
    * 2 Light sedation; briefly awakens to voice (eye opening/contant) < 10 seconds
    * 3 Moderate sedation; movement or eye opening. No eye contact
    * 4 Deep sedation; no response to voice, but movement or eye opening to physical stimulation
    * 5 Unarousable; no response to voice or physical stimulation

SECONDARY OUTCOMES:
mean arterial pressure | Before induction ,After intubation 1 min,After intubation 5 min, After intubation 15 min After intubation 30 min
  mmHg
Heart rate | Before induction ,After intubation 1 min,After intubation 5 min, After intubation 15 min After intubation 30 min
  beats/min

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, Kayapınar, Turkey (Türkiye)